CLINICAL TRIAL: NCT06585059
Title: A Phase Ib Clinical Study of TQB2928 in Combination With a Third-Generation EGFR TKI in Patients With Advanced Non-Small Cell Lung Cancers
Brief Title: Clinical Trial of TQB2928 in Combination With a Third-Generation Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor (TKI) in Patients With Advanced Non-Small Cell Lung Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2928-Ib-03
Record Dates: First submitted 2024-09-01; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-06

CONDITIONS: Advanced Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2928 injection + Almonertinib Mesilate Tablets (Experimental): Every 3 weeks constitutes one treatment cycle. For the first 2 cycles, TQB2928 is administered via infusion once a week. Starting from the 3rd cycle, TQB2928 is administered once every 3 weeks. Amivantamab is taken orally at a fixed time daily.
  Interventions: Drug: TQB2928 injection + Almonertinib Mesilate Tablets

INTERVENTIONS:
Drug: TQB2928 injection + Almonertinib Mesilate Tablets — TQB2928 is a recombinant fully humanized Immunoglobulin G4 (IgG4) monoclonal antibody that can promote tumor cell phagocytosis by macrophages and exert anti-tumor effects.
  Almonertinib Mesilate Tablets is a third generation of EGFR-TKI targeting drug.

SUMMARY:
This is a Phase Ib study to evaluate the safety, tolerability, and efficacy of TQB2928 in combination with third-generation EGFR TKIs in subjects with advanced non-small cell lung cancer, and to determine the recommended Phase II dose (RP2CD).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years; Eastern Cooperative Oncology Group (ECOG) score: 0-1; Expected survival of more than 3 months；
* Locally advanced or metastatic NSCLC diagnosed by histology or cytology
* The major organs are functioning well；
* Negative serum pregnancy test within 7 days prior to the first dose and must be a non-lactating subject, female and male subjects of childbearing potential should agree to use contraception for the duration of the study and for 6 months after the end of the study；
* Subjects voluntarily joined this study, signed the informed consent form, and had good compliance.

Exclusion Criteria:

* Current concomitant presence of other malignancies within 5 years prior to the first dose;
* Unresolved toxicity above CTCAE Grade 1 due to any prior anti-tumor therapy;
* Significant surgical treatment, biopsy, or significant traumatic injury within 28 days prior to the first dose;
* Long-term unhealed wounds or fractures;
* Cerebrovascular accident (including transient ischemic attack, intracerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism within 6 months prior to the first dose;
* A history of psychotropic drug abuse and cannot be abstained from or have a mental disorder;
* Subjects with any severe and/or uncontrolled disease;
* History of live attenuated vaccination within 2 weeks prior to the first dose or planned live attenuated vaccination during the study;
* Previous history of unexplained severe allergies, hypersensitivity to monoclonal antibodies or exogenous human immunoglobulins, or hypersensitivity to TQB2928 injection or excipients in pharmaceutical formulations;
* According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patients or affect the completion of the study, or subjects who are considered to be unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase II recommended combination doses (RP2CD) | Baseline up to 24 months
  The recommended dosage for drug combination therapy in the second phase of clinical trials (i.e. Phase II clinical trials).
Objective Response Rate (ORR) | Up to 2 years
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria.
Duration of Response (DOR) | Up to 2 years
  Defined as the time from first documented response to documented disease progression.
Progression-free survival (PFS) | Up to 2 years
  Defined as the time from the first dose of TQB2928 to the first occurrence of disease progression or death from any cause.
Time to Progression | Up to 2 years
  The time from randomization to obtaining the first objective relief.

SECONDARY OUTCOMES:
Elimination half-life (t1/2) | Cycle 1 Day1: in 0.5 hour pre-dose and immediately after dose, 2, 6, 24 hours; Day1 and Day15 of Cycle 1, Cycle 2 Day1: in 0.5 hour pre-dose and immediately after dose; Day1 on Cycle 3, Cycle 4, Cycle 5: in 0.5 hour pre-dose (each cycle is 3 weeks)
  The time required for plasma drug concentration to decrease by half.
Area under the plasma concentration-time curve (AUC0-last) | Cycle 1 Day1: in 0.5 hour pre-dose and immediately after dose, 2, 6, 24 hours; Day1 and Day15 of Cycle 1, Cycle 2 Day1: in 0.5 hour pre-dose and immediately after dose; Day1 on Cycle 3, Cycle 4, Cycle 5: in 0.5 hour pre-dose (each cycle is 3 weeks)
  The area enclosed by the plasma concentration curve against the timeline.
Apparent Plasma Clearance (CL) | Cycle 1 Day1: in 0.5 hour pre-dose and immediately after dose, 2, 6, 24 hours; Day1 and Day15 of Cycle 1, Cycle 2 Day1: in 0.5 hour pre-dose and immediately after dose; Day1 on Cycle 3, Cycle 4, Cycle 5: in 0.5 hour pre-dose (each cycle is 3 weeks)
  Apparent plasma clearance of TQB2928.
Apparent volume of distribution(Vz) | Cycle 1 Day1: in 0.5 hour pre-dose and immediately after dose, 2, 6, 24 hours; Day1 and Day15 of Cycle 1, Cycle 2 Day1: in 0.5 hour pre-dose and immediately after dose; Day1 on Cycle 3, Cycle 4, Cycle 5: in 0.5 hour pre-dose (each cycle is 3 weeks)
  The ratio of the amount of TQB2928 in the body to the blood concentration.
Steady-state trough concentration (Css-min) | Cycle 1 Day1: in 0.5 hour pre-dose and immediately after dose, 2, 6, 24 hours; Day1 and Day15 of Cycle 1, Cycle 2 Day1: in 0.5 hour pre-dose and immediately after dose; Day1 on Cycle 3, Cycle 4, Cycle 5: in 0.5 hour pre-dose (each cycle is 3 weeks)
  Minimum concentration during dosing.
Immunogenicity: anti-drug antibody (ADA) | From the time of informed consent signed through 90 days after the last dose
  Incidence of anti-drug antibody (ADA).
Adverse Events (AE) rate | From date of the first dose until the date of 30 days after last dose or new anti-tumor treatment, whichever came first
  The occurrence and severity of all AEs.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China